CLINICAL TRIAL: NCT06423430
Title: Treatment ResistAnt Depression Subcallosal CingulatE Network DBS
Brief Title: Treatment ResistAnt Depression Subcallosal CingulatE Network DBS (TRANSCEND)
Acronym: TRANSCEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABT-CIP-10494
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Treatment Resistant Depression
Keywords: DBS; Major Depressive Disorder; Bilateral Stimulation; Antidepressant Treatment; neurostimulation; ABT-CIP-10494
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham-stimulation group (Sham Comparator): Group will be implanted with DBS system but device is not activated for the first 12 months. After 12 months, this group can receive stimulation.
  Interventions: Device: Sham-stimulation
- Active-stimulation group (Active Comparator): Group will have DBS system activated 2 weeks post-implant.
  Interventions: Device: Active-stimulation

INTERVENTIONS:
Device: Sham-stimulation — Sham-stimulation
  Arms: Sham-stimulation group
Device: Active-stimulation — Active DBS
  Arms: Active-stimulation group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of bilateral stimulation of the subcallosal cingulate white matter (SCCwm) using Deep Brain Stimulation (DBS) as an adjunctive treatment of non-psychotic unipolar Major Depressive Disorder (MDD) in adults.

DETAILED DESCRIPTION:
The aim of this prospective, multi-centered, double-blind, randomized, delayed-stimulation/ Sham-stimulation controlled 12-month study is to evaluate the effectiveness and safety of bilateral stimulation of the subcallosal cingulate white matter (SCCwm) using the Infinity™ Deep Brain Stimulation (DBS) system as an adjunctive treatment of non-psychotic unipolar Major Depressive Disorder (MDD) for adults who are experiencing a Major Depressive Episode (MDE) with inadequate response to 4 or more antidepressant treatments.

In a double-blind fashion, half the subjects will receive active DBS therapy, while half will receive sham stimulation. After the 12-month endpoint, all subjects will be unblinded to their treatment group, and subjects in the control arm will receive active DBS therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be diagnosed with non-psychotic unipolar Major Depressive Disorder.
2. The patient must be in a major depressive episode for ≥12 months or have had at least 3 lifetime depressive episodes.
3. The patient has tried and failed a minimum of four different types of antidepressant treatments as measured by a tool designed for this purpose.
4. Depression medication and treatment regimen must be stable for a minimum of 4 weeks before the first baseline visit

Exclusion Criteria:

1. Pregnant or those who plan to become pregnant during study
2. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that could limit participation in the study or interfere with adherence to the study protocol.
3. Current or lifetime history of psychotic features in any Major Depressive Episode.
4. Has an intracranial Central Nervous System disease that impairs motor, sensory or cognitive function or that requires intermittent or chronic medication.
5. Significant acute suicide risk.
6. Diagnosis of Substance Use Disorder or Alcohol Use Disorder without sustained remission (12 months or longer).
7. Current and ongoing use of neurostimulation treatment that may interfere with DBS therapy/system.
8. Treatment with another investigational device or investigational drugs.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS total score | 12 months
  The MADRS absolute change is measured as score change from baseline to the endpoint evaluation period.
  The Montgomery Asberg Depression Rating Scale (MADRS) consists of 10 items, and each item is rated on a 7-point Likert scale. The sum of the item scores produces a MADRS total score that ranges from 0 to 60, with higher scores reflecting greater depression severity.
CGI-I response rate | 12 months
  The CGI-I response is defined as a rating of "very much improved" or "much improved." The Clinical Global Impression of Severity and Improvement (CGI-I) is a clinician-rated tool used to measure the global impression of a treatment response in a patient's by comparing their baseline condition (i.e., before DBS system implant) with their current state.

SECONDARY OUTCOMES:
Percent time in MADRS response | 12 Months
  The Montgomery Asberg Depression Rating Scale (MADRS) consists of 10 items, and each item is rated on a 7-point Likert scale. The sum of the item scores produces a MADRS total score that ranges from 0 to 60, with higher scores reflecting greater depression severity.
Percent time in MADRS partial response | 12 Months
  The Montgomery Asberg Depression Rating Scale (MADRS) consists of 10 items, and each item is rated on a 7-point Likert scale. The sum of the item scores produces a MADRS total score that ranges from 0 to 60, with higher scores reflecting greater depression severity.
Percent time in CGI-I partial response | 12 Months
  The Clinical Global Impression of Severity and Improvement (CGI-I) is a clinician-rated tool used to measure the global impression of a treatment response in a patient's by comparing their baseline condition (i.e., before DBS system implant) with their current state.
MADRS Response Rate | 12 Months
  The Montgomery Asberg Depression Rating Scale (MADRS) consists of 10 items, and each item is rated on a 7-point Likert scale. The sum of the item scores produces a MADRS total score that ranges from 0 to 60, with higher scores reflecting greater depression severity.
Q-LES-Q score change | 12 Months
  The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-report measure that assess the degree of enjoyment and satisfaction experienced by patients in various areas of daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kopell, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Mark George, MD, Principal Investigator — Medical University of South Carolina
Locations (24):
- United States (24):
  - University of Alabama at Birmingham - Dept. of Psychiatry, Birmingham, Alabama
  - USC University Hospital, Los Angeles, California
  - UCLA Department of Psychiatry, Los Angeles, California
  - University of California at Davis, Sacramento, California
  - USF Health, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Mount Sinai Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Med. Ctr, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No